CLINICAL TRIAL: NCT02980497
Title: Determination of the Antiplaque/Antigingivitis Efficacy of Essential Oil Containing Mouthrinses In a Six-Month Study
Brief Title: Antiplaque/Antigingivitis Efficacy of Essential Oil Mouthrinses in Six-Month Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Collaborators: University of Taubate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FCLGBP0056
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Plaque; Gingivitis; Gum Inflammation; Bleeding
Keywords: mouthrinse; plaque; gingivitis; gum bleeding
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis; Hemorrhage; Gingival Hemorrhage | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Listerine Zero Mouthwash (without alcohol) (Active Comparator): Brushing twice daily in the usual manner with an ADA-Accepted Fluoride Toothpaste (Colgate Cavity Protection) using a soft-bristled toothbrush and rinsing with 20 ml of Listerine Zero Mouthwash (without alcohol) for 30 seconds.
  Interventions: Other: Listerine Zero Mouthwash (without alcohol)
- Listerine Antiseptic Mouthwash (with alcohol) (Active Comparator): Brushing twice daily in the usual manner with an ADA-Accepted Fluoride Toothpaste (Colgate Cavity Protection) using a soft-bristled toothbrush and rinsing with 20 ml of Listerine Antiseptic Mouthwash (with alcohol) for 30 seconds.
  Interventions: Other: Listerine Antiseptic Mouthwash (with alcohol)
- Brush only (No Intervention): Brush only twice daily in the usual manner with an ADA-Accepted Fluoride Toothpaste (Colgate Cavity Protection) using a soft-bristled toothbrush.

INTERVENTIONS:
Other: Listerine Zero Mouthwash (without alcohol) — 20 ml of rinse for 30 seconds, twice a day
  Arms: Listerine Zero Mouthwash (without alcohol)
Other: Listerine Antiseptic Mouthwash (with alcohol) — 20 ml of rinse for 30 seconds, twice a day
  Arms: Listerine Antiseptic Mouthwash (with alcohol)

SUMMARY:
The objective of this randomized, single-center, examiner-blind, controlled, parallel group, six-month clinical study is to compare the antiplaque/antigingivitis potential of a no-alcohol essential oil containing mouthrinse and an alcohol essential oil containing mouthrinse. A negative control group using only an ADA Accepted anticavity toothpaste will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older, in good general and oral health, except gingivitis.
2. Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon research site personnel's assessment;
3. Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial.
4. A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count.
5. A mean gingival index ≥ 1.75 according to the Modified Gingival Index.
6. A mean plaque index ≥ 1.95 according to the Turesky modification of the Quigley-Hein Plaque Index scored on six surfaces per tooth.
7. Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator.
8. Absence of moderate/advanced periodontitis based on a clinical examination (ADA Type III, IV).
9. Absence of fixed or removable orthodontic appliance or removable partial dentures.

Exclusion Criteria:

1. History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes and mouthrinses and red food dye.
2. History of serious medical conditions that, at the discretion of the Investigator, will disqualify the subject.
3. History of rheumatic fever, heart murmur, mitral valve prolapse or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures.
4. Antibiotic, anti-inflammatory or anticoagulant therapy during the study or within the 2 weeks prior to the baseline exam.
5. Regular use of chemotherapeutic antiplaque/antigingivitis products such as triclosan, essential oil, cetylpyridinium chloride, or chlorhexidine containing mouthrinses within the 2 weeks prior to baseline.
6. Current or history of alcohol or drug abuse.
7. Self reported pregnancy or lactation (this is an exclusion criterion due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Mean Modified Gingival Index (MGI) at 6 Months | 6 Months
  Gingivitis was assessed on the buccal and lingual marginal gingivae and interdental papillae on all scoreable teeth on a 5-grade categorical scale of 0=normal to 4=severe inflammation.

SECONDARY OUTCOMES:
Mean Modified Gingival Index (MGI) at 1 Month | 1 Month
  Gingivitis was assessed on the buccal and lingual marginal gingivae and interdental papillae on all scoreable teeth on a 5-grade categorical scale of 0=normal to 4=severe inflammation.
Mean Modified Gingival Index (MGI) at 3 Months | 3 Months
  Gingivitis was assessed on the buccal and lingual marginal gingivae and interdental papillae on all scoreable teeth on a 5-grade categorical scale of 0=normal to 4=severe inflammation.
Mean Gingival Bleeding Index (BI) at 1 Month | 1 Month
  Gingival bleeding was assessed at four gingival areas (distobuccal, mid-buccal, mid-lingual, and mesiolingual) around each tooth on a 3-grade categorical scale of 0=absence of bleeding after 30 seconds, 1=bleeding after 30 seconds, and 2=immediate bleeding.
Mean Gingival Bleeding Index (BI) at 3 Months | 3 Months
  Gingival bleeding was assessed at four gingival areas (distobuccal, mid-buccal, mid-lingual, and mesiolingual) around each tooth on a 3-grade categorical scale of 0=absence of bleeding after 30 seconds, 1=bleeding after 30 seconds, and 2=immediate bleeding.
Mean Gingival Bleeding Index (BI) at 6 Months | 6 Months
  Gingival bleeding was assessed at four gingival areas (distobuccal, mid-buccal, mid-lingual, and mesiolingual) around each tooth on a 3-grade categorical scale of 0=absence of bleeding after 30 seconds, 1=bleeding after 30 seconds, and 2=immediate bleeding.
Mean Plaque Index (PI) (Turesky Modification of the Quigley Hein PI) at 1 Month | 1 Month
  Plaque area was scored on six surfaces (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) of all scorable teeth on a 6-grade categorical scale of 0=no plaque to 5=plaque covering 2/3 or more of the surface.
Mean Plaque Index (PI) (Turesky Modification of the Quigley Hein PI) at 3 Months | 3 Months
  Plaque area was scored on six surfaces (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) of all scorable teeth on a 6-grade categorical scale of 0=no plaque to 5=plaque covering 2/3 or more of the surface.
Mean Plaque Index (PI) (Turesky Modification of the Quigley Hein PI) at 6 Months | 6 Months
  Plaque area was scored on six surfaces (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) of all scorable teeth on a 6-grade categorical scale of 0=no plaque to 5=plaque covering 2/3 or more of the surface.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cortelli, Ph. D, Principal Investigator — Universidade de Taubate; Sheila Cortelli, Ph.D, Study Chair — Universidade de Taubate
Locations (1):
- University of Taubate, Taubaté, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lynch MC, Cortelli SC, McGuire JA, Zhang J, Ricci-Nittel D, Mordas CJ, Aquino DR, Cortelli JR. The effects of essential oil mouthrinses with or without alcohol on plaque and gingivitis: a randomized controlled clinical study. BMC Oral Health. 2018 Jan 10;18(1):6. doi: 10.1186/s12903-017-0454-6. PMID 29321067